CLINICAL TRIAL: NCT07196046
Title: A Randomized Double-Blind, Comparator-Controlled, Single-Site Study With a Single-Blind Placebo Run-In and Crossover Design to Evaluate Joint Comfort in Adults Using Enhanced Bioavailability Curcumin Dietary Supplements
Brief Title: Product Responsiveness to Enhanced Bioavailability Curcumin Dietary Supplements in Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ultra Botanica LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: UBL-2024
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Joint Discomfort; Quality of Life (QOL)
MeSH Terms: interventions — TARGET 1 dietary supplement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Supplement order will vary based on randomization.
  Interventions: Dietary Supplement: Supplement 2; Dietary Supplement: Supplement 3; Dietary Supplement: Supplement 1
- B (Experimental): Supplement order will vary based on randomization.
  Interventions: Dietary Supplement: Supplement 2; Dietary Supplement: Supplement 3; Dietary Supplement: Supplement 1

INTERVENTIONS:
Dietary Supplement: Supplement 2 — A dietary supplement administered daily for 30 days. This supplement is being evaluated as part of a randomized, double-blind, crossover study to assess its effect on joint comfort. This product may be a placebo.
Dietary Supplement: Supplement 3 — A third dietary supplement administered daily for 30 days. This supplement is being evaluated as part of a randomized, double-blind, crossover study to assess its effect on joint comfort. This product may be a placebo.
Dietary Supplement: Supplement 1 — A dietary supplement administered daily for 14 days. This supplement is being evaluated as part of a randomized, double-blind, crossover study to assess its effect on joint comfort. This product may be a placebo.

SUMMARY:
The goal of this clinical trial is to evaluate whether two distinct formulations of bioavailable curcumin supplements can improve joint comfort in adults who experience self-reported discomfort. Participants will also receive a placebo during the study, but they will not know when they receive it.

The main questions it aims to answer are:

* Do participants report improved joint comfort after taking each curcumin-based supplement?
* Are there difference in quality-of-life scores or pain perceptions between the two products?

Researchers will compare the effects of two different formulations of bioavailable curcumin supplements to see if one provides greater improvements in joint comfort and related outcomes.

Participants will:

* Wear a fitness tracker starting at the time of electronic consent to provide continuous data on physical activity, heart rate, and sleep
* Take two supplements twice daily for 30 days, then complete a 7-day break (washout), followed by 30 days on the second supplement
* Take one supplement twice daily for 14 days then complete a 7-day break (washout)
* Complete validated questionnaires throughout the study to report on joint comfort, quality of life, and overall health
* Participate in a 30-day follow up period after the final supplement to complete final questionnaires and wearable data collection

The study is conducted remotely using the Alethios decentralized research platform.

ELIGIBILITY:
Inclusion Criteria

1. Able to provide a digital or wet signed informed consent to participate in the study
2. Willing and able to comply with all study requirements and instructions of the site study staff
3. Meets the study inclusionary criteria and voluntarily gives informed consent for participation
4. Male or female, 30 to 85 years old (inclusive)
5. Ambulatory without use of a walker or cane
6. Study participant must be symptomatic (self-professed, not diagnosed) for 6 months or longer
7. Occasional mild to moderate discomfort and/or pain of major or collection of minor joints defined by a level of 4-8 on screening NRS
8. No known clinically significant liver abnormality (e.g. cirrhosis, transplant, etc.).
9. Possession of a functional wearable device (e.g., Apple Watch, Fitbit, Garmin) compatible with the Alethios platform and willingness to link it to the platform for continuous data collection during the study period, and able to use the device for the study duration.

Exclusion Criteria

1. A history of allergic reactions to Dairy or Dairy proteins, Turmeric, or Curcumin
2. Any medical history of joint disease or pain syndrome interfering with evaluation of joint discomfort, such as rheumatoid arthritis, psoriatic arthritis, gout, aseptic necrosis, joint replacement, complex regional pain syndrome, fibromyalgia, peripheral neuropathy, or malignancy (left to Principal Investigator (PI) discretion)
3. Presence of significant medical, neurological, or psychiatric condition that could interfere with ambulation or self-assessment ability such as: unmanaged diabetes, uncontrolled hypertension, heart failure, Alzheimer's disease, Parkinson's disease, intracranial hemorrhage, multiple sclerosis, or traumatic brain injury (left to Principal Investigator (PI) discretion)
4. Liver, kidney, gallbladder, or peptic ulcer disease, or active disorders of the intestinal tract that may interfere with supplement absorption, distribution, or clearance.
5. Surgery, hospitalization, or fracture within the 6 months prior to screening.
6. Presence of discomfort and/or pain that in a self-professed description severely limits mobility.
7. Any pharmacological or non-pharmacological treatment targeting joint discomfort that was initiated or modified within 4 weeks prior to randomization
8. Prohibited Medications & Treatments - The following medications and treatments are not permitted during the study: a. Intra-articular (IA) injections of any kind; b. Blood thinners; c. Opioid-containing analgesics; d. Topical treatments targeting joint discomfort; e. Systemic medical treatments that may interfere with liver or kidney function or ambulation; f. Immunosuppressants; g. Corticosteroids exceeding 5 mg prednisone equivalent per day (If ≤5 mg prednisone, the dose must be stable for at least 6 months.); h. Non-steroidal anti-inflammatory drugs (NSAIDs) such as ibuprofen or naproxen
9. Regular consumption of >7 standard alcoholic drinks/week where 1 standard drink is 0.6 fluid ounces of "pure" ethanol and is equivalent to 12 oz of beer (5% alc/vol), 5 oz wine (12% alc/vol), or 1.5 oz distilled spirits (40% alc/vol).
10. Pregnant or breastfeeding individuals will be excluded from participation due to the lack of safety data on these formulations in these populations. Participants who become pregnant during the study must notify the study team immediately and will be withdrawn from the study.
11. As a result of the medical review and screening investigation, the Principal Investigator considers the study participant not suitable for the study due to limitations in self-assessment ability, difficulty with ambulation, conditions interfering with perception of joint discomfort, or conditions or medications that preclude safe use of supplement.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Quality-of-Life Scores (RAND-36) | Onboarding, Day 32, Day 69, Day 98
  Change in RAND-36 scores across the eight domains (physical functioning, role limitations, pain, general health, vitality, social functioning, emotional well-being, and mental health). Scores will be compared within and across supplement phases to evaluate participant-perceived quality of life.

SECONDARY OUTCOMES:
Self-Reported Joint Comfort (PGI-Style Scales) | Day 2, Day 8, Day 15, Day 21, Day 29, Day 39, Day 46, Day 53, Day 58, Day 66, Day 69, Day 98
  Participant-reported changes in joint comfort and general well-being using PGI-style scales. Instruments ask participants to compare their current experience to baseline using a 7-point global impression scale.
Pain and Discomfort Ratings (NRS) | Day 2, Day 8, Day 15, Day 21, Day 29, Day 39, Day 46, Day 53, Day 58, Day 66, Day 69, Day 98
  Numeric Rating Scale (NRS)
Timing of Perceived Impact | Day 2 through Day 69
  Participant-reported timing of initial improvement in joint comfort following the start of each supplement phase. Captured through structured response options (e.g., within hours, day)
Rescue Medication Use | Day 8, Day 15, Day 21, Day 29, Day 46, Day 53, Day 58, Day 66
  Participant reports of rescue pain medication use (e.g., ibuprofen, acetaminophen), including frequency and perceived effectiveness
Supplement Compliance | Day 8, Day 15, Day 21, Day 29, Day 46, Day 53, Day 58, Day 66
  Self-reported adherence to the prescribed supplement intake schedule. Includes reasons for missed doses.

OTHER OUTCOMES:
Wearable-Derived Activity and Sleep Metrics | From eConsent to study completion; data collected before starting any intervention and then collected weekly
  Continuous collection of step count, heart rate variability, and sleep duration using a wearable device. Used for exploratory correlations with self-reported comfort and quality-of-life outcomes
End-of-Phase Supplement Reflections | Day 32 and Day 69
  Participant summaries of their experiences during each supplement phase, including joint comfort, mobility, and alignment with expectations. Includes multiple-choice and optional open-text responses

CONTACTS AND LOCATIONS:
Overall Officials: Adam Payne, CEO, MBA, Principal Investigator — Ultra Botanica LLC
Locations (1):
- Ultra Botanica LLC, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided
The Sponsor has not yet determined whether individual participant data (IPD) from this study will be shared. Given the small sample size and potential risk of re-identification, a decision will be made after study completion and data analysis.

REFERENCES:
- See also: MAPI Research Trust. (n.d.). Patient Global Impressions scale - Change, Improvement, Severity (PGI-C, PGI-I, PGI-S) (eProvide, Ed.) [Review of Patient Global Impressions scale - Change, Improvement, Severity (PGI-C, PGI-I, PGI-S)] — https://eprovide.mapi-trust.org/instruments/patient-global-impressions-scale-change-improvement-severity